CLINICAL TRIAL: NCT05786300
Title: Is Early Superimposed Neuromuscular Electrical Stimulation (NMES+) Useful to Improve Muscle Tissue Recovery From Type 3a/3b Hamstring Strain Injuries (HSI)?
Brief Title: Effect of NMES+ on Hamstring Lesion (3a/3b)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università degli studi di Roma Foro Italico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMESHAMSTRING1
Record Dates: First submitted 2023-03-01; First posted 2023-03-27 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Hamstring Injury; Muscle Rupture; Hamstring Sprain
Keywords: Electrical Muscle Stimulation (EMS); NMES+; Hamstring strain injury; Neuromuscular Electrical Stimulation (NMES)
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): The Treatment Group will follow the rehabilitation protocol with the addition of the Neuromuscular Electrical Stimulation Superimposed onto Movement (NMES+) as part of the rehabilitation protocol.
  1st/2nd Week at 35 Hertz. 3rd/4th Week 50 Hertz. 5th/6th Week 70 Hertz
  Interventions: Device: NMES+; Procedure: Rehab
- Control Group (Active Comparator): The Control Group will follow the same rehabilitation protocol with no addition of the NMES+.
  A weight-bearing protocol with a week by week progression on load, repetitions and sets.
  Interventions: Procedure: Rehab

INTERVENTIONS:
Device: NMES+ — The Treatment Group will follow the rehabilitation protocol with the addition of the NMES+.
  1st/2nd Week at 35 Hertz. 3rd/4th Week 50 Hertz. 5th/6th Week 70 Hertz.
  Arms: Treatment Group
Procedure: Rehab — The Control Group will follow a protocol based on the latest available guidelines for the rehabilitation of the hamstrings lesions.
  A weight-bearing protocol with a week by week progression on load, repetitions and sets.

SUMMARY:
The goal of this clinical trial is to analyze the effect of the electrical stimulation superimposed onto movement in healthy semi-professional athletes who sustained a type 3a/3b hamstring strain injury.

The main questions it aims to answer are:

* Is NMES+ useful for the treatment of type 3a/3b hamstring strain injury?
* Does NMES+ improve the quality of the injured muscle tissue? Participants will follow a 3 week protocol, following the latest evidence available.[describe the main tasks participants will be asked to do, treatments they'll be given and use bullets if it is more than 2 items]. If there is a comparison group: Researchers will compare [insert groups] to see if [insert effects].

ELIGIBILITY:
Inclusion Criteria:

* recreational or semi-professional athletes
* Body Mass Index between 18,5 e 24,9
* Hamstring strain lesion type 3a/3b

Exclusion Criteria:

* previous hamstring strain lesions
* Anterior Cruciate Ligament Reconstruction using Hamstring graft
* Current hamstring strains

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Tear monitoring and muscle quality | Baseline
  Healing status of the muscle tear (mm/cm), using ultrasounds
Tear Monitoring | Up to 6 weeks
  Healing status of the muscle tear (mm/cm), using ultrasounds